CLINICAL TRIAL: NCT06883942
Title: Pilot Study on the Evaluation of the Functionality, Safety and Reliability of New Tripping Devices for Lower Limbs.
Acronym: MOTU++ pedane
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Biorobotic Institute Scuola Superiore sant'Anna Pisa (Unknown)
Responsible Party: Sponsor
Other Study IDs: MOTU++ Studio Clinico Pedane
Record Dates: First submitted 2025-02-14; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Lower Limb Amputation; Slip Perturbations; Fall Risk
Keywords: amputation; stumble; slipping; lower limb; fall risk

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with unilateral trans-femoral and/or trans-tibial amputation.
  Interventions: Procedure: prosthetic group performs the entire protocol with their own prosthesis; Device: Experimental Group

INTERVENTIONS:
Procedure: prosthetic group performs the entire protocol with their own prosthesis — The 1st session is the enrolment and functional evaluation one. The following 2 we test the algorithm functionality verification; one session for both platforms. The last 2 sessions are necessary to acquire prognostic markers for falls; one session for both platforms.
  The balance disturbance tests will take place on two platforms:
  * The sliding platform consists of a metal supporting structure and a wooden cover, which has a manual release mechanism that allows the activation of the tile responsible for simulating the events that occur during sliding.
  * The stumbling platform consists of a metal supporting structure and a wooden cover, which features an electronically activated plastic and foam tripping mechanism that simulates the sequence of events that occur during a stumble.
Device: Experimental Group — The fall detection algorithm will be evaluated first. In a second step, the experimentally obtained prognostic markers of fall risk will be studied. The markers thus obtained shall be validated by comparison with markers already established in clinical practice or in the literature.

SUMMARY:
The study aims to identify prognostic biomarkers of fall risk in patients with lower limb amputation

DETAILED DESCRIPTION:
The protocol will involve both trans-tibial and trans-femoral amputation subjects, for a total duration of up to 5 sessions.

Initially, the fall detection algorithm will be evaluated on trans-femoral and trans-tibial amputees performing the test while wearing their prosthesis.

In a second step, the experimentally obtained prognostic markers of fall risk will be studied (i.e., using one or both of the perturbation platforms described below).

The markers thus obtained are to be validated by comparison with markers already established in clinical practice or in the literature.

Experimental platforms The platforms are composed of a mechanism to simulate and investigate the aid that the prosthetic system can provide in the event of a source of tripping and/or slipping.

ELIGIBILITY:
Inclusion Criteria:

* Trans-femoral or trans-tibial lower limb amputation;
* Functional medical classification: Level K3-K4;
* Subjects who have had a prosthesis for at least 1 year (experienced wearers);
* Informed consent signed by the subject

Exclusion Criteria:

* Significant medical comorbidities (severe neurological disease, cardiovascular disease diabetes/unstabilised hypertension, severe sensory deficits);
* Cardiac device wearers (PMK or AICD);
* Cognitive impairment (MMSE adjusted for age and schooling <24);
* Inability or unwillingness to provide informed consent;
* Severe depressive symptomatology - Beck Depression Inventory (BDI-II <19);
* Severe anxiety symptoms - State-Trait Anxiety Inventory (STAI-Y <50).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects with monolateral trans-femoral and/or trans-tibial.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
algorithm validation | baseline
  Verifying the measurement performance of the trip and slip detection algorithm on prosthesis wearers

SECONDARY OUTCOMES:
data aquiring | baseline
  Acquire data on amputees to be used for the development of a new version of the detection algorithm and its testing.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang F, D'Andrea SE, Nunnery MJ, Kay SM, Huang H. Towards design of a stumble detection system for artificial legs. IEEE Trans Neural Syst Rehabil Eng. 2011 Oct;19(5):567-77. doi: 10.1109/TNSRE.2011.2161888. Epub 2011 Aug 18. PMID 21859635
- [Result] Palumbo P, Randi P, Moscato S, Davalli A, Chiari L. Degree of Safety Against Falls Provided by 4 Different Prosthetic Knee Types in People With Transfemoral Amputation: A Retrospective Observational Study. Phys Ther. 2022 Apr 1;102(4):pzab310. doi: 10.1093/ptj/pzab310. PMID 35079822
- [Result] Hunter SW, Batchelor F, Hill KD, Hill AM, Mackintosh S, Payne M. Risk Factors for Falls in People With a Lower Limb Amputation: A Systematic Review. PM R. 2017 Feb;9(2):170-180.e1. doi: 10.1016/j.pmrj.2016.07.531. Epub 2016 Jul 30. PMID 27485674
- [Result] Miller WC, Speechley M, Deathe B. The prevalence and risk factors of falling and fear of falling among lower extremity amputees. Arch Phys Med Rehabil. 2001 Aug;82(8):1031-7. doi: 10.1053/apmr.2001.24295. PMID 11494181